CLINICAL TRIAL: NCT06846281
Title: A Randomized, Open-label, Parallel-group, Non-inferiority Study Comparing Efficacy, Safety, and Tolerability of Remibrutinib After Switching From Ocrelizumab in Participants Living With Relapsing Multiple Sclerosis, Followed by Open-label Treatment With Remibrutinib
Brief Title: Efficacy and Safety of Remibrutinib After Switching From Ocrelizumab in Participants Living With Relapsing Multiple Sclerosis.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLOU064C12306; 2023-509275-17 (Other: EU CTIS)
Record Dates: First submitted 2025-02-24; First posted 2025-02-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: MS; RMS; Remibrutinib; LOU064; Ocrelizumab; Age; MRI; T2 lesions; NEDA-3
MeSH Terms: interventions — remibrutinib; ocrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Remibrutinib Core (Experimental): Remibrutinib tablet taken orally
  Interventions: Drug: Remibrutinib oral treatment
- Ocrelizumab Core (Active Comparator): Ocrelizumab at standard dose and route of administration (i.v. or s.c) per label
  Interventions: Drug: Ocrelizumab
- Remibrutinib Extension (Experimental): Remibrutinib tablet taken orally
  Interventions: Drug: Remibrutinib oral treatment
- Remibrutinib Extension (Ocrelizumab in Core) (Experimental): Remibrutinib tablet taken orally
  Interventions: Drug: Remibrutinib oral treatment

INTERVENTIONS:
Drug: Remibrutinib oral treatment — Remibrutinib tablet taken daily
  Other Names: LOU064
  Arms: Remibrutinib Core; Remibrutinib Extension; Remibrutinib Extension (Ocrelizumab in Core)
Drug: Ocrelizumab — Ocrelizumab 600mg infusion or 920mg injection
  Arms: Ocrelizumab Core

SUMMARY:
The purpose of this Phase 3b study is to assess the efficacy, safety and tolerability of remibrutinib after switching from ocrelizumab and compared to continuous ocrelizumab treatment, in patients living with relapsing multiple sclerosis (plwRMS).

DETAILED DESCRIPTION:
The study is a randomized, open-label, non-inferiority multi-center, Phase 3b study to provide efficacy, safety, and tolerability data for remibrutinib after switching from ocrelizumab and in comparison to continuous ocrelizumab in plwRMS.

This study consists of an initial Core Part (CP) (maximum duration per participant of up to 24 months), followed by an Extension Part (EP) (of up to 24 months duration) for eligible participants.

All participants completing the 24-month treatment of the Core Part of the study may be eligible to continue in the Extension Part, an open-label, single-arm, fixed-dose design in which participants are treated with remibrutinib for up to 24 months.

The study will be conducted in the USA among other countries globally.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female aged 40 to 70 years (inclusive)
* Diagnosis of RMS according to the 2017 McDonald diagnostic criteria
* Treated with ocrelizumab according to routine clinical practice and at standard dose
* Neurologically stable within 30 days
* Suitable to be switched to remibrutinib based on physician judgement or patient preference

Key Exclusion Criteria:

* Diagnosis of primary progressive multiple sclerosis (PPMS) according to the revised 2017 McDonald criteria
* History of clinically significant Central Nervous System disease or neurological disorders
* History of confirmed Progressive Multifocal Leukoencephalopathy or neurological symptoms consistent
* Active clinically significant systemic bacterial, viral, parasitic or fungal infections
* Active, chronic disease of the immune system other than MS
* Severe cardiac disease or significant findings on the ECG
* Participant who is unable to undergo MRI scans
* History of life-threatening infusion or injection reaction related to ocrelizumab

Other inclusion and exclusion criteria may apply

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2030-01-30 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of new or enlarging T2 lesions_Core Part | Baseline up to month 24
  Number of new/enlarging T2 lesions per year on MRI at month 24 (relative to baseline)

SECONDARY OUTCOMES:
Participants with no evidence of disease activity-3 (NEDA-3)_Core Part | Baseline up to month 24
  Participants with no evidence of disease activity-3 (NEDA-3), as assessed by absence of confirmed MS relapses, 6-month confirmed disability progression (6mCDP) and new/enlarging T2 lesions on MRI
Number of adverse events (AEs) and serious adverse events (SAEs)_Core Part | Baseline up to month 24
  Adverse events will be collected throughout the trial. Any safety assessment findings such as laboratory, vital signs, electrocardiogram data that are considered clinically significant or meet the protocol definition of an adverse event will be reported as adverse event or serious adverse event, as appropriate
Annualized rate of new or enlarging T2 lesions_Extension Part | Month 24 up to month 48
  Number of new/enlarging T2 lesions per year on MRI
Participants with no evidence of disease activity-3 (NEDA-3)_Extension Part | Month 24 up to month 48
  Participants with no evidence of disease activity-3 (NEDA-3), as assessed by absence of confirmed MS relapses, 6-month confirmed disability progression (6mCDP) and new/enlarging T2 lesions on MRI
Number of Adverse events and serious adverse events_Extension Part | Month 24 up to month 48
  Adverse events will be collected throughout the trial. Any safety assessment findings such as laboratory, vital signs, electrocardiogram data that are considered clinically significant or meet the protocol definition of an adverse event will be reported as adverse event or serious adverse event, as appropriate

CONTACTS AND LOCATIONS:
Locations (69):
- United States (16):
  - Perseverance Research Center, Scottsdale, Arizona
  - Neurology of Central FL Res Ctr, Altamonte Springs, Florida
  - University of Florida, Gainesville, Florida
  - Neurology Associates PA, Maitland, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - University of Kansas Hospital, Kansas City, Kansas
  - Michigan Institute of Neurological, Farmington Hills, Michigan
  - Memorial HC Ins for Neuroscience, Owosso, Michigan
  - Holy Name Medical Center, Teaneck, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Sanford Health, Fargo, North Dakota
  - Premier Neurology, Greenville, South Carolina
  - Sibyl Wray MD Neurology PC, Knoxville, Tennessee
  - Austin Regional Clinic, Austin, Texas
  - John Peter Smith Hospital, Fort Worth, Texas
- Argentina (2):
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Buenos Aires
- Australia (4):
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, St Leonards
- Novartis Investigative Site, Bruges, Belgium
- Canada (3):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Lévis, Quebec
  - Novartis Investigative Site, Montreal, Quebec
- Denmark (2):
  - Novartis Investigative Site, Aarhus N
  - Novartis Investigative Site, Glostrup Municipality
- France (10):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
- Greece (3):
  - Novartis Investigative Site, Chaïdári
  - Novartis Investigative Site, Larissa
  - Novartis Investigative Site, Thessaloniki
- Italy (6):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
- Mexico (2):
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Mexico City
- Portugal (3):
  - Novartis Investigative Site, Braga
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
- Slovakia (2):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Trnava
- South Africa (2):
  - Novartis Investigative Site, Cape Town, Western Cape
  - Novartis Investigative Site, Pretoria
- Spain (9):
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Switzerland (3):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- Novartis Investigative Site, Swansea, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.